CLINICAL TRIAL: NCT07263087
Title: Health Profile of the Elderly Population in a Rural Area of Assiut Governorate: A Community-Based Cross-Sectional Study
Brief Title: Elderly Health Profile in a Rural Village of Assiut
Acronym: RURAL-AGE
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Galal Eldeen Abdelhamid, Assistant Lecturer of Public Health & Community Medicine, Assiut University
Other Study IDs: PHCM-ElderlyHealth-2025-ASSIUT
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Diseases in Older Adults; Malnutrition; Frailty; Functional Decline Geriatric Health
Keywords: Elderly Health; Geriatric Assessment; Nutrition in Older Adults; Functional Status; Chronic Disease Burden; Rural Health; Upper Egypt
MeSH Terms: conditions — Malnutrition; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults (≥60 Years): Community-dwelling older adults aged 60 years and above living in Al-Boura village, Assiut, Egypt. Participants will complete structured interviews and undergo basic anthropometric and clinical assessments. No interventions are provided as this is an observational, cross-sectional study.

SUMMARY:
This study aims to assess the health, nutrition, functional status, and quality of life of older adults living in Al-Boura village in Assiut, Egypt. It is an observational, community-based study that includes adults aged 60 years and above. Participants will complete interviews covering medical history, lifestyle behaviors, functional ability, mental health, nutrition, and quality of life. Physical measurements such as weight, height, blood pressure, and simple clinical assessments will also be performed. The goal of the study is to describe the current health needs of the elderly population and identify risk factors for chronic diseases, malnutrition, and functional decline. The results will help guide local health services and future elderly-care programs in Upper Egypt. No treatments or interventions will be given as part of this study.

DETAILED DESCRIPTION:
This community-based observational study aims to provide a comprehensive assessment of the health status, nutritional profile, functional ability, mental health, and quality of life of older adults residing in Al-Boura village in Assiut, Upper Egypt. The study is designed to describe the current health needs of individuals aged 60 years and above through structured interviews, standardized assessment tools, and objective anthropometric and clinical measurements.

Participants will be evaluated using validated instruments covering chronic disease history, medication use, health behaviors, activities of daily living (ADLs), instrumental activities of daily living (IADLs), cognitive status, depression, frailty, nutritional risk, and quality of life. Physical examinations will include measurements such as weight, height, body mass index (BMI), blood pressure, mid-upper arm circumference, and waist circumference. The study does not involve any interventions, randomization, or treatment allocation.

The primary objective is to identify the prevalence of chronic conditions, malnutrition, functional decline, frailty, and psychosocial challenges among the elderly population in rural settings. Secondary objectives include identifying associated factors, mapping unmet health needs, and generating evidence to support planning and implementation of elderly-focused health programs in Upper Egypt. Findings from this study are expected to guide the development of community health strategies and inform future public health interventions aimed at improving elderly care and reducing disease burden in resource-limited rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Resident in the selected rural village in Assiut
* Able to communicate and respond to interview questions
* Provides informed consent to participate

Exclusion Criteria:

* Bedridden or severely ill preventing participation
* Severe cognitive impairment preventing interview
* Refusal to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes elderly individuals aged 60 years and older residing in Al-Boura village, Assiut Governorate. Participants are recruited directly from households using systematic random sampling. Both men and women from all socioeconomic backgrounds are eligible.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Geriatric Health Problems | At baseline (single assessment at time of interview)
  Proportion of older adults (≥60 years) identified with one or more geriatric health problems assessed during the study visit, including chronic diseases (hypertension, diabetes), functional limitation, cognitive impairment, malnutrition risk, depression, polypharmacy, and sensory impairment. These assessments are conducted through structured questionnaires, anthropometric measurements, and clinical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital - Public Health and Community Medicine Department, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
o. The study will not share individual participant data (IPD) because the dataset contains sensitive personal health information from elderly participants in a small rural community. Public sharing of raw individual-level data may compromise participant confidentiality and privacy. Only aggregated, de-identified results will be reported in publications."